CLINICAL TRIAL: NCT02341053
Title: Effects of Standing on Non-Ambulatory Children With Spinal Muscular Atrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gillette Children's Specialty Healthcare (Other)
Collaborators: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1411M55281
Record Dates: First submitted 2015-01-02; First posted 2015-01-19 (Estimated); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Spinal Muscular Dystrophy; Neuromuscular Disability
Keywords: SMA; Neuromuscular disability

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Load-measuring platform (Other): Load-sensing platform A load-sensing platform will be placed under each foot of the subject to record the time course of load borne by each of the lower extremities during weight-bearing training in an assisted standing device.
  Intervention: Assisted Standing Treatment Program. Assisted standing treatment program will gradually increase their duration of standing by up to 75% after the baseline phase.
  Interventions: Other: Assisted Standing Treatment Program

INTERVENTIONS:
Other: Assisted Standing Treatment Program — Assisted Standing Treatment Program - Assisted standing treatment program will be gradually increase duration of standing by up to 75% after baseline.

SUMMARY:
Non-ambulatory children with a neuromuscular disability such as spinal muscular atrophy (SMA) are at significant risk for poor bone health as defined by low bone mineral density (BMD) and increased propensity to fracture. Poor bone health is thought to be related, at least in part, to abnormally low levels of load experienced by the skeleton. A common physical approach for increasing bone density is to stimulate the musculoskeletal system by increasing the amount and duration of weight-bearing in the lower extremities. For non-ambulatory individuals, this takes the form of using an assisted standing device to enable the child to spend time in a standing position with some degree of weight placed on the lower limbs. Some of these physical interventions demonstrate variable improvement in BMD in children with neuromuscular conditions, and some do not. A serious limitation in the previous work in this area is a failure to objectively measure the magnitude and duration of the loading experienced by the lower extremities. Thus, a lack of change in BMD may be due to the extremities experiencing only a fraction of the body weight (due to load-sharing with the assistive device) for an inadequate duration of standing time.

In order to investigate the efficacy of standing treatment for increasing BMD, the investigators will develop a simple, portable and inexpensive transducer that will measure the magnitude and time course of the load experienced by the lower extremities of individuals with SMA who use a stationary assisted standing device. The specific goal of this proposed project will be to develop, validate and establish the initial feasibility of such a measurement device.

DETAILED DESCRIPTION:
Background: Non-ambulatory children with a neuromuscular disability such as spinal muscular atrophy (SMA) are at significant risk for poor bone health as defined by low bone mineral density (BMD) and increased propensity to fracture. Poor bone health is thought to be related, at least in part, to abnormally low levels of load experienced by the skeleton. A common physical approach for increasing bone density is to stimulate the musculoskeletal system by increasing the amount and duration of weight-bearing in the lower extremities. For non-ambulatory individuals, this takes the form of using an assisted standing device to enable the child to spend time in a standing position with some degree of weight placed on the lower limbs. Some of these physical interventions demonstrate variable improvement in BMD in children with neuromuscular conditions, and some do not. A serious limitation in the previous work in this area is a failure to objectively measure the magnitude and duration of the loading experienced by the lower extremities. Thus, a lack of change in BMD may be due to the extremities experiencing only a fraction of the body weight (due to load-sharing with the assistive device) for an inadequate duration of standing time.

Methods: In order to investigate the efficacy of standing treatment for increasing BMD, we will develop a simple, portable and inexpensive transducer that will measure the magnitude and time course of the load experienced by the lower extremities of individuals with SMA who use a stationary assisted standing device. This transducer will consist of an array of sensors embedded within a mat that will be placed under an individual's feet while they are in assisted standing. A prototype will be validated by comparing the output of this load-sensing mat against known loads that will be applied to the surface of the mat statically. The specific characteristics of the loading in the lower extremities of subjects can then be correlated with changes in their BMD to obtain a true outcome assessment. As a demonstration of this approach, we will recruit 3 children with SMA from Gillette Children's Specialty Healthcare who are currently participating in a standing program. Once enrolled and informed consent is obtained, the participants will use the mat provided to them to collect load and duration data during a baseline period where they will continue their standing program, and during a subsequent intervention period where they will increase the duration of their standing. The specific goal of this proposed project will be to develop, validate and establish the initial feasibility of such a measurement device.

Implications: Successful completion of this proposed project will provide the necessary groundwork to move forward with a multicenter clinical trial on a large number of subjects with a variety of neuromuscular conditions. The measurement device will allow us to correlate change in BMD with the specific load history for each participant, thereby allowing us to determine whether physical interventions can lead to increased BMD in individuals with neuromuscular disabilities. Analysis of the data will help define a dose-dependent relationship between load, duration and changes in BMD, thereby guiding providers and therapists in prescribing standing interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Age 3-14 years old
2. Diagnosed with Spinal Muscular Atrophy (SMA)
3. Participating in a standing program using a stationary assisted standing device.
4. Gross Motor Function Classification System (GMFCS) Level IV or V
5. Parent must be able to provide consent.

Exclusion Criteria:

1. Currently on bisphosphonates

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2016-09-08 (Actual); Primary Completion 2018-07-25 (Actual); Study Completion 2018-07-25 (Actual)

PRIMARY OUTCOMES:
Collection of load magnitude and duration data (Use load-sensing platforms to collect load magnitude and duration during standing treatment program) | 12 months
  Use load-sensing platforms to collect load magnitude and duration during standing treatment program.

SECONDARY OUTCOMES:
Bone Mineral Density | 12 months
  Determine whether an increase in the duration of standing leads to improvements in BMD, fracture incidence, pulmonary function and quality of life, and whether there is evidence that relationships exist between these outcome measures and load magnitude and duration.

CONTACTS AND LOCATIONS:
Overall Officials: Walter Truong, MD, Principal Investigator — Gillette Children's Specialty Healthcare
Locations (1):
- Gillette Children's Specialty Healthcare, Saint Paul, Minnesota, United States